CLINICAL TRIAL: NCT06254625
Title: Fecal Transplantation in Patients With Colonic Diverticulitis: a Pilot Study
Brief Title: Fecal Transplantation in Patients Colonic Diverticulitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Bjørsum-Meyer, Principal investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 333-2023-AK
Record Dates: First submitted 2023-12-04; First posted 2024-02-12 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Diverticulitis, Colonic; Colon Inflamed
Keywords: Fecal microbiome; Fecal microbiome transplantation; Colonic diverticulitis
MeSH Terms: conditions — Diverticulitis, Colonic; Colitis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiome transplantation (Experimental): 25-30 capsules are ingested with apple juice or coca cola light, and the patient is observed for 30-60 minutes before they are allowed to go home. The capsules are to be ingested within 4 hours of thawing. Each transplant, comprising 25-30 capsules, contain 50 g of feces originating from one donor.
  Interventions: Other: Fecal Microbiome
- Placebo (Placebo Comparator): The placebo group receives 25-30 placebo capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fecal Microbiome — Fecal microbiome transplantation from a healthy donor.
  Arms: Fecal microbiome transplantation
Other: Placebo — Place capsules
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the safety and effect of fecal microbiome transplantation (FMT) in patients with a former episode of acute colonic diverticulitis. The main question[s] it aims to answer are:

* Is FMT in patients with a former episode of acute colonic diverticulitis a safe procedure without severe adverse events
* What is the impact of FMT on patient-reported outcomes and re-admission rate

Participants will be asked to:

* to ingest either 25-30 capsules with FMT or placebo capsules
* Fill-in GI-QLI questionnaire prior to treatment/placebo and 3 months post baseline
* Fill-in eating habit questionnaire
* deliver blood-and stool samples prior to treatment/placebo and 3 months post baseline
* In both the treatment and placebo group 5 patients will be offered sigmoideoscopy for mucosal biopsies if it is more than 2 items]. If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects]

DETAILED DESCRIPTION:
Colon diverticulosis (CD) is a prevalent condition, and its global incidence appears to be rising due to the aging population and an increasing number of younger individuals affected. Symptoms may encompass abdominal pain, changes in bowel habits, and bloating. The prevailing hypothesis suggests that CD arises from chronic constipation, resulting in heightened intraluminal pressure, colonic muscular hypertrophy, and mucosal herniation. However, the etiology remains incompletely understood, involving complex interactions among genetic factors, gut microbiota, and diet. The path from CD to diverticulitis is believed to involve diverticular obstruction, alterations in the gut microbiome, local tissue ischemia, and micro-perforations. Recent studies provide evidence supporting the role of altered colonic microbiota in CD pathogenesis, showing compositional changes in the microbiome of inpatients with acute diverticulitis (AD) characterized by decreased diversity and abundance of commensal microbiota as compared to healthy controls.

Traditionally, diverticulitis has been treated with antibiotics due to its association with bacterial overgrowth in the large intestine. However, prolonged antibiotic therapy has led to complications, such as Clostridioides difficile infection (CDI). Currently, studies are exploring the clinical evidence supporting the use of antibiotics for uncomplicated diverticulitis.

Fecal microbiota transplantation (FMT) has emerged as a novel therapeutic approach for recurrent CDI, involving the transfer of stool from healthy donors to the gastrointestinal tract of a recipient/patient. FMT is considered a safe and effective strategy to restore a healthy diversity of the gastrointestinal microbiota in patients with CDI. Furthermore, systematic reviews have demonstrated positive responses of FMT in managing inflammatory bowel disease (IBD), showcasing local therapeutic immune-modulating abilities.

Typically, patients with AD present with acute pain, tenderness in the left lower quadrant, fever, and elevated infection parameters. AD severity is categorized as uncomplicated diverticulitis or complicated diverticulitis, using the Hinchey classification. In Denmark, the diagnosis of diverticulitis is confirmed with a CT scan during acute hospitalization. While optical colonoscopy (OC) is rarely used for diagnostic purposes in the clinical setting due to the risk of complications, patients are offered a follow-up OC after conservative AD treatment, typically six weeks after inflammation resolution, to exclude malignancy.

Purpose The investigators aim to evaluate clinical and patient-reported efficacy, safety, and impact on the colonic microbiome of one FMT or one placebo-FMT administered via capsules in patients with diverticulitis.

Study Design The study is designed as a randomized controlled trial (RCT) with the primary objective of investigating the feasibility, tolerability and safety of FMT in patients with acute uncomplicated diverticulitis at Odense University Hospital (Odense/Svendborg).

Patient selection: The study population will consist of patients admitted to Odense University Hospital Patients with acute uncomplicated diverticulitis. Eligible patients will be identified during hospital admission and assessed for inclusion in the study. To be eligible, the diverticulitis in the patient must be acute uncomplicated, as confirmed by CT scan. After hospital discharge, eligible patients will be offered the opportunity to participate in the study.

Informed Consent: All prospective participants will be required to provide both verbal and written informed consent before they are included in the study. Invitees will also be informed that they have the option to decline FMT treatment at the day of capsule administration. If the patient chooses to refuse participation, they will be offered no further treatment, as planned at hospital discharge.

Sample Size and Randomization: The study will include a total of 40 patients, all of whom have CT-confirmed diverticulitis. These patients will be randomized 1:1 into two study arms.

* Active Treatment Group: This group will comprise 20 patients who will receive FMT in capsule form.
* Control Group: The control group will also consist of 20 patients who will receive placebo treatment also in capsule form.

Blinding: The study will be conducted in a double-blind manner to minimize bias. Neither the personnel nor the patients will be aware of whether FMT is administered or not in the capsules. A designated coordinator will coordinate with clinical immunological department, which will then deliver the products, along with the transplantation journal (whether FMT or placebo), to the core department of the patients.

In summary, this study employs a RCT design to assess the feasibility, tolerability, and safety of FMT in patients with acute uncomplicated diverticulitis. A total of 40 patients will be enrolled and randomly assigned to either the active treatment group (FMT) or the control group (placebo). The study will be blinded to ensure impartial evaluation of outcomes. Eligible patients will provide informed consent before participating in the study.

Endpoints

* Primary efficacy endpoint: Proportion of patients treated with antibiotics within 3 months following FMT comparing FMT and placebo.
* Primary safety endpoint: Patient safety monitored by a) number of re-admissions, and b) number of adverse events within 3 months of FMT.
* Secondary endpoints: Change from baseline to 3 months in the GI-QLI questionnaire. Change from baseline to 3 months in: fecal bacteria composition and metabolism; intestinal permeability (measured by specific markers in plasma); plasma and fecal calprotectin; specific circulating inflammatory markers (ie, cytokines, adipokines and chemokines); and macroscopic and microscopic inflammatory changes of the colonic mucosa.

Recruitment of patients The recruitment of patients will occur within the Surgical Department or Emergency department at Odense University Hospital (Odense/Svendborg). Patient enrollment takes place during hospital admission in conjunction with their acute diverticulitis episode. The first contact with the patients is initiated by the attending physician following a CT scan confirming uncomplicated diverticulitis and when the patient's condition stabilizes with conservative treatment.

Upon informing the patient that they have uncomplicated diverticulitis and do not need or will get any further treatment, the attending doctor will also provide information about the project, including an explanation of FMT is and its former use. Subsequently, the attending doctor will make a referral to either Camilla Thorndal Nielsen or Thomas Bjørsum-Meyer, who will then contact the patient to provide verbal information with the aim of facilitating enrollment during the hospital stay. In cases where the patient has not been informed during admission, a meeting will be offered 14 days after discharge. Furthermore, the patients will have the opportunity to undergo a sigmoidoscopy, the primary purpose of which is to obtain biopsies for examination of the colonic mucosa. This will be performed at baseline (prior to FMT administration) and at 3 months after. To consent to this, there will be a checkbox to mark on the consent form.

Patients will be informed about the right for the presence of a layman representative during discussions and their right to a period of reflection within an undisturbed room prior to making a decision regarding participation. Furthermore, patients will be presented with the option of physical or online follow-up consultation with either Thomas Bjørsum-Meyer or Camilla Thorndal Nielsen, scheduled for 14 days after discharge. To ensure clarity, patients will be provided with the pamphlets titled "Forsøgspersoners rettigheder i et sundhedsvidenskabeligt forskningsprojekt" and "Før du besluttter dig", as well as our Participant Information on the trial. Written consent will be obtained prior to the patient's discharge. Alternatively, patients may provide written consent for participation during the consultation scheduled 14 days after discharge. Failure to receive a response from a patient regarding their participation within 14 days following hospital discharge, will render them ineligible for participation.

The Study Procedure At the out-patient consultation 14 days after hospital discharge the patients will receive a fecal sampling and be instructed to fill 3-5 fecal samples. If the patient has consented to the sigmoidoscopy they will be instructed to fill the fecal samples BEFORE they start the regimen of bowel cleansing. Before the FMT procedure they will be asked to fill in 2 questionnaires to report on their symptoms: the Eating Habits Questionnaire and the Gastrointestinal Quality of Life (GI-QLI). Both questionnaires will be sent in a digital mail via e-boks or by mail. The GI-QLI is a 36-item multidimensional scale covering symptoms, and physical, emotional, and social dysfunction relating to gastrointestinal diseases or their treatments. It is an appropriate and validated tool to assess health-related quality of life in clinical studies in patients with gastrointestinal disease. Each of the 36 items are scored on a 5-point Likert scale and summed to get overall GI-QLI score. The Eating Habits questionnaire covers the patient's average eating habits in the last month.

At the day FMT treatment, they will bring the fecal samples to the clinic. In the clinic on the day of the FMT treatment they will have blood samples taken. The intervention will be conducted at the patient's core department: the surgical department at Odense University Hospital (Odense/Svendborg/Nyborg). If they have agreed to a sigmoidoscopy, there will be taken brush biopsies of the mucosa, in both the treatment group and the placebo group.

Three months post baseline the patients will receive the QI-GLI questionnaire digitally again, as well as another fecal sampling set by mail, which they will be asked to bring when they have their blood samples taken for the second time and, for those it may be relevant undergo the second sigmoidoscopy.

The investigators will monitor and report safety outcomes by re-admissions, adverse events and need for antibiotics, during the whole study period.

Randomization The randomization will be managed by randomization tool in Open REDCap. The patients, care providers, and outcome assessors will remain unaware of the group assignments, and only de-identified codes will be used to link participants to their data during the study to maintain their confidentiality. In case of exceptional circumstances when knowledge of the treatment allocation is essential for further management of the patient, the trial secretary will reveal the assigned intervention to the treating doctor. However, patients, trial care providers and outcome assessors will remain blinded as far as possible. Cases of unblinding will be registered and reported. The study will be terminated when 40 patients have been included in total, which is anticipated to be achieved within a 6-months period.

The FMT procedure Use of capsule-based fecal microbiota transplantation has been shown to be clinically effective approach to restore intestinal microbiota composition and is now the preferred form of administration. This non-invasive oral delivery provides an easy route of administration and a newfound flexibility for clinicans and patients. 25-30 capsules are ingested with apple juice or coca cola light, and the patient is observed for 30-60 minutes before they are allowed to go home. The capsules are to be ingested within 4 hours of thawing. Each transplant, comprising 25-30 capsules, contain 50 g of feces originating from one donor. The placebo group receives placebo capsules. The patients will only receive the FMT or placebo capsules once.

Collecting of biological material Fecal samples: The patient will collect 5 stool samples consisting of 1g each. The same material for biobanking will be collected at both baseline and 3 months follow-up. The investigators will investigate the fecal microbioal composition (i.e, bacteria, virus, fungi, and archea) and microbial activity using metagenomics/16S, culturomics, proteomics, and metabolomis. Fecal samples will also be taken if the patient is admitted in need for antibiotics, prior to the treatment.

Blood samples: At baseline the patient will have 5 blood tests taken, and this will again be done at the 3 months follow-up. Markers of intestinal permeability will be investigated such as plasma zonulin, zonulin-related protein, calprotectin, I-FABP, CD14, and LPS. Furthermore, Analyses of inflammation-related plasma proteins using the Olink 92 inflammation panel (link) or a similar protein assay will be conducted.

Brush biopsy: During the baseline sigmoidoscopy and the second one, a brush biopsy (0.1g / 1x1 mm) will be obtained from the gastrointestinal mucosa of the patient's colon. The purpose of this procedure is to examine the microenvironment in the diverticula, focusing on inflammation or other microbiological abnormalities. Both paraffin-fixed tissue for immunohistochemistry and tissue stored in RNALater for proteomics will be collected.

All brush biopsies, blood samples and fecal samples will be stored in a research biobank for current and future research with the subject's consent. Four biobanks (A, B, C and D) will be established:

A. Blood samples biobanking (both patients and donors)

- 5 x Plasma-EDTA 1 ml (2.0 ml Sarstedt tubes)

B. Fecal samples biobanking (patients)

* 5 x 1 g stool from each donation
* 1 x brush biopsy of gastrointestinal mucosa (0.1 g / 1x1 mm)

C. Screening samples (donor)

* 2 x 7 blood samples (4 ml)
* 2 x 1 fecal sample (15 g)
* 2 x 1 urine sample (5 ml)
* 5 x swab SARS CoV2 PCR test

D. Fecal samples biobanking (donors)

* 3 x 1 g stool from each donation
* 3 x 1 g FMT transplant from each donation

At the end of the project, any additional material will continue to be stored in their respective biobanks, for future research, if the subjects consent to this.

Recruitment of donors The recruitment of donors will occur at the Blood bank at Odense University Hospital, Stærmosegårdsvej 6, 5230 Odense M. Donors will be sourced from active members of the Danish blood donor corps. The recruitment of stool donors will take place through discussions and material exchanges with the Blood Bank personnel during their blood donations appointments.

When donors express interest in the project, comprehensive verbal information about the project is provided by a medical doctor affiliated the Blood Bank. Donors are made aware that they have the option to bring a layperson representative and are entitled to a period of reflection. In additions, they will be encouraged to read the pamphlets titled "Forsøgspersoners rettigheder i et sundhedsvidenskabeligt forskningsprojekt" and "Før du besluttter dig". The reflection period, starting from the conveyance of verbal information and extending to the procurement of informed consent, will span 1 week. Subsequently, our written participant information document will be provided to the selected donors.

Stool donors: The stool donor corps will consist of 2 anonymous (to the recipient) donors who must be healthy as assessed by screening questionnaire and be active members of the Danish blood donor corps, age 25-55 years, body mass index between 18.5 and 25 kg/m2 and an average alcohol intake <7 (women) and <14 (men) units per week. No alcohol intake within a week of donation is allowed, and no systemic medication including antibiotics and NSAIDs 6 months prior to the donation are allowed. The donor must eat a balanced diet (no extreme low-calorie or high-calorie diets) and must not be in a stressful life period. Before joining the stool donor corps, each potential donor will go through a screening process including stool analyses for fecal calprotectin and enteric pathogens (Aeromonas, Campylobacter, C. difficile, diarrhoeagenic Escherichia coli, Salmonella, Shigella, Vibrio, Yersinia enterocolitica and multidrug-resistant bacteria), parasites including microscopy of ova and cysts, Entamoeba histolytica/dispar (DNA), Cryptosporidium (DNA) and Giardia (DNA), sapo-virus (RNA), rotavirus (RNA), human astrovirus (RNA), human adenoviruses (DNA) and noroviruses (RNA), a Helicobacter pylori antigen test, blood test for CRP) (acceptable level: <6.0 mg/L), white blood cell count (acceptable range: 3.50-8.8x10^9/L), hemoglobin (acceptable range: 8.3-10.5 mmol/L), albumin (acceptable range: 36-50g/L), alanine aminotransferase (acceptable range:10-70 U/L), estimated glomerular filtration rate (acceptable range:>59 mL/min) and coeliac disease, and blood test for infectious agents including current infection with Epstein-Barr virus (IgM) and cytomegalovirus (IgM), hepatitis A, B, C and E, tuberculosis (QuantiFERON TB-Gold test), syphilis, HIV (ab HTLV1/2), E. histolytica (antibodies) and Strongyloides (antibodies), and a urine test for Chlamydia Trachomatis and Neisseria gonorrhoeae (DNA/RNA). After passing the screening tests, the donor will donate stool for the next month after which, the donor will have to pass the screening program once more before the stool can be released for transplantation.

Preparing the FMT suspension: Donors will collect stool at home and transport it in a cooling bag to the study within 1 hour. Stool will be sieved to remove particulate material, followed by dilution in sterile saline (0.9% NaCl) and 10% glycerol, The FMT suspension will be stored at -80 degree C until use. On the day of the FMT transplantation, the transplant suspension (250 mL) will be thawed to 37degree C and subsequently apportioned into five 50 mL syringes. When preparing the final FMT solution, it's sought to split pools from the same batch, however if there are less than five splits remaining from the same donation date, it is allowed to split from the same donor collected on different dates. The optimal storage life for frozen stool product has yet to be clarified, but it is widely accepted that the transplant material can be stored at -80 degree C for 2 years, and most likely much longer.

Information from patient files Departments including patients will contact the investigator and co-investigator, when they find a patient, which they deem suitable for the study. The investigator and co-investigator will then approach these patients, with information about the project.

Information that is extracted before consent to participate and forwarded to the researcher:

* Personal registration number (CPR)
* Age
* Gender
* Earlier hospitalization, especially with diverticulitis
* Earlier treatment with antibiotics within 12 months prior to inclusion
* Comorbidities and diseases, and other, which could be reason for exclusion.
* CT findings
* Symptoms at admission with acute diverticulitis

Information that is extracted after consent to participate, which gives project manager, sponsors and sponsor represents, as well as control authorities direct access to obtain information in patient journals.

* Symptoms after discharge (if any)
* Intake of antibiotics
* Readmission
* Patient file on sigmoidoscopy procedure.
* Symptoms and possible readmission after treatment
* Patient reported earlier antibiotic use. Data is used if patients' needs to be excluded while the project is running.

Management of patient information in the project Data on participants will be collected from electronic patient files and questionnaires. Only relevant information for conducting the study is extracted. Data will be entered via a secure web-based electronic clinical report form into a central RedCap database hosted by Odense Patient data Explorative Network at Odense University Hospital. Data obtained during the clinical examination will be entered directly into the database. Also, patient questionnaires will be filled out directly into the database. Access to the study data will be restricted, and a password system will be used to control access. All information about the patients' health and other private matters is covered by confidentiality, as well as information about biobank materials. The information will continue to be so after the project ends, this also includes material that will continue to be stored in one of the research biobanks. Gathered information on participants is protected according to the "Legislation on the Processing of Personal Data" and "Danish Health Care Act". The authorization from Danish Data Protection Agency will be secured.

Risks and side effects The treatment that is being offered here, is identical with the treatment that is given as routine to patients with CDI. It is the same product, amount of the product and procedure. This has run routinely at Odense University Hospital for the last 5 years since 2017. The most frequently reported short-term minor adverse events (AEs) related to FMT are vomiting, mild diarrhea, abdominal cramping, transient fever, and elevated CRP. The possible serious short-term AE's related to the procedure are rare and primarily not related to the administration of FMT. These include complications of the endoscopy, such as perforation and bleeding, and complications related to the sedation, such as aspiration.

A recent systematic review has investigated the adverse events of FMT and found a total incidence rate of 28.5%, in 50 relevant studies with a total of 1089 patients. In 5 out of 42 publications the events were definitely related to the FMT procedure, but in the remaining 38 they were described as probably related. The most common FMT AE was abdominal discomfort and reported in 19 publications. The incidences of serious adverse events (SAEs) for FMT were 2.0% and 6.1% for upper and lower gastrointestinal routes, respectively. The SAEs that possibly were related to FMT included infections (0.7%), IBD flare (0.6%), death (0.3%), autoimmune disease and FMT procedure-related injury.

Although most of the knowledge on FMT related AEs are from patients who have suffered from CDI and/or IBD, these findings request caution when performing FMT. However, FMT is in general considered safe, especially with a strict screening of donors, and even elderly patients with poor medical condition as well as immunosuppressed patients have been proven to tolerate the procedure well.

In the present study, the investigators will carefully monitor and evaluate safety by means of open assessment of adverse events. All reported or observed adverse events are recorded by the investigators and will be monitored until resolution, stabilization or until it has been shown that the study intervention is not the cause. The National Cancer Institute Common Terminology Criteria for Adverse Events V.4.03 (NIH publication #09-7473) will be used to grade the severity of AEs. Gastrointestinal side effects (nausea, vomiting, abdominal pain, number of stools per week, stool type (Bristol Stool Chart) blood or mucus in stool) will be registered by the patients once a week for the first month following the randomized intervention. Subject incidence rates of all treatment-emergent AEs will be tabulated by system organ class and preferred term. Tables of fatal AEs, severe AEs, AEs leading to withdrawal from study and significant treatment-emergent AEs, will also be provided.

Statistical considerations When designing this trial, no prior data for FMT efficacy in patients with diverticulitis were available. However, the investigators found it reasonable to assume that if patients with acute uncomplicated diverticulitis should be willing to receive FMT as a future standardized treatment, the procedure should at least provide an effect size well beyond a moderate effect size. A smaller group of patients has been chosen, since this is a pilot study, and it is not known how the patients with diverticulitis will respond to the treatment with FMT.

Statistical methods The full analysis set will consist of all randomized participants, which will be analyzed according to their randomized treatment group, so the participants allocated to a treatment group will be followed up, assessed, and analyzed as members of that group, irrespective of their compliance to the planned treatment (intention-to-treat principle). The safety analysis set will include all patients who were randomly assigned to a study group and has exposure to a transplant (independent of group). Descriptive statistics will be provided for demographics and baseline characteristics. The summary statistics of continuous variables will include N, mean, SD, median, interquartile range and range. All summaries presenting frequencies and incidences will include counts, percentages, and the total number of participants in the corresponding arm.

Ethics and dissemination This study is designed as a proof-of-concept clinical trial and will be performed in agreement with Good Clinical Practice (GCP) standards, and in accordance with the ethical standards of the responsible committee on human experimentation (institutional and national) and with the Helsinki Declaration (64th, 2013). The trial will be started after the regional ethics committee and the Data Protection Agency has approved the protocol. Data will be handled according to the General Data Protection Regulation (GDPR) and the Data Protection Act.

The Danish Health and Medicines Authority does not classify the FMT procedure as a medical intervention and has had no objection to the use of FMT for this study and patient category. Thus, no GCP auditing is legally required. A report describing any potential side effects and AEs will be submitted to the Ethics Committee yearly. Suspected Unexpected Serious Adverse Reactions will be reported to the Ethics Committee within 7 days. Based on these reports, the Ethics committee can determine to terminate the trial early. The Danish Patient Compensation Association provides compensations for patients injured in connection to medical clinical trials. Although the Danish Health Authorities, for the time being, do not classify donor fecal microbiota as tissue, all steps of the stool donor recruitment, stool donation and FMT preparation will be in accordance with the Danish Tissue Law to ensure that the quality and safety standards laid down in the Danish Legislation BEK nr 764 of 26 May 2015 (implementing Directive 2004/23/EC) are met. Stool donors will be recruited from the South Danish Transfusion Service & Tissue Centre, Department of Clinical Immunology, Odense University Hospital, and they will be carefully screened for potentially transmissible infections and other conditions associated with gut microbiota function before their stool can be released for FMT. Being a stool donor is voluntary, and no compensation fee will be given. Furthermore, to ensure donor traceability, each patient in the active treatment arm will only receive microbiota from one donor. Also, frozen stool products will be clearly labelled with a unique donation code based on the ISBT 128 coding and labelling system, and the release of the final product will adhere to the standards for tissue and blood donation.

Due to uncomplicated diverticulitis being a common disease, with no treatment with great clinical evidence, the identification of new treatment modalities is essential to help the physician. All patients with acute uncomplicated diverticulitis, who are participating in this study, would not receive any treatment, and therefore the patient population would benefit greatly from new treatment options. The trial will be registered at ClinicalTrials.gov, and important protocol modifications will be updated here. Dissemination will occur through publications in international peer-reviewed journal(s). Positive as well as negative results will be published. The investigators plan to publish the clinical findings (primary and secondary endpoints) in one publication with CN as first author and TB as last author. The tertiary endpoints will be published separately in one or more publications.

Economics Initiative for the study was taken by Thomas Bjørsum-Meyer. The costs of the study will be covered by OUH, Region of Southern Denmark and external funds. No funds have yet been granted or applied for. The grants will cover the costs of establishing and maintaining the 4 research biobanks, practical costs (i.e. mail services), secretary, as well as the costs of blood samples, stool samples and colonic mucosa biopsies and the FMT procedure. The Trial Manager has no financial affiliation with study subjects or other interests in the study. Funding is administered by an account subject to public audit.

ELIGIBILITY:
Inclusion Criteria:

- CT-confirmed Acute Uncomplicated Diverticulitis: Eligible patients should have a confirmed diagnosis of acute uncomplicated diverticulitis based on in-hospital CT scans.

The condition must be defined as an infection limited to the colon, not extending to the peritoneum, and the patients should not require antibiotics treatment for their diverticulitis.

This definition ensures that the study focuses on cases of uncomplicated diverticulitis.

- Admission to Odense University Hospital (Odense/Svendborg): Participants must be admitted to Odense University Hospital in Odense or Svendborg for the diagnosis and initial management of acute uncomplicated diverticulitis

Exclusion Criteria:

* Inability to provide Informed Consent: Patient who are unable to comprehend the study information and provide informed consent due to cognitive impairment, language barriers or any other reason will be excluded.
* Cognitive or Physical Impairment: Patients with disabilities that hinder their ability to comply with the study procedures, either cognitively or physically, will be excluded.
* Complicated Diverticulitis: patients with complicated diverticulitis, as defined by the presence of abscesses, fistulas, perforations, or other severe complications on the CT scan, will not be eligible for participation.
* CT Findings Requiring Biopsy or Polyp Removal: Individuals with CT findings indicating the need for colonoscopy to perform biopsy (e.g., suspected cancer) or for polyp removal will not be eligible for the study.
* Presence of Other Gastrointestinal Diseases: Patients with other gastrointestinal diseases, for such as IBD, will be excluded to maintain a homogeneous study population.
* Immunocompromised Patients: Individuals with known immunodeficiency disorders or undergoing immunosuppressive thearapy will be excluded due to potential safety concerns associated with FMT.
* Impaired Renal Function: Patients with impaired renal function may be more susceptible to potential risks or complications associated with experimental intervention, and their inclusions could confound the results or increase the likelihood of adverse evenets.
* History of FMT: Patients with a previous history of FMT will be excluded rom the study to avoid any potential confounding factors.
* Pregnant and Lactation: Pregnant or lactating individuals will not be included to ensure the safety of both the mother and the fetus/infant..
* Allergies to Active Substances in the Trial: Patients with known allergies to the active substances administered in the trial will not be eligible for participation.
* Participation in Other Clinical Trials: Individuals currently participating in other clinical trials involving investigational drugs or interventions will not be eligible to avoid potential interference with study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients treated with antibiotics within 3 months following FMT comparing FMT and placebo. | 3 months
Patient safety monitored by a) number of re-admissions, and b) number of adverse events within 3 months of FMT. | 3 months

SECONDARY OUTCOMES:
Change from baseline to 3 months in the GI-QLI questionnaire | 3 months
Change from baseline to 3 months in: fecal bacteria composition and metabolism | 3 months
  Changes in intestinal permeability (measured by specific markers in plasma); plasma and fecal calprotectin; specific circulating inflammatory markers (ie, cytokines, adipokines and chemokines); and macroscopic and microscopic inflammatory changes of the colonic mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bjørsum-meyer, M.D., PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Funen, Denmark

REFERENCES:
- [Derived] Thorndal C, Kragsnaes MS, Nilsson AC, Holm DK, dePont Christensen R, Ellingsen T, Kjeldsen J, Bjorsum-Meyer T. Safety and efficacy of faecal microbiota transplantation in patients with acute uncomplicated diverticulitis: study protocol for a randomised placebo-controlled trial. Therap Adv Gastroenterol. 2025 Jan 2;18:17562848241309868. doi: 10.1177/17562848241309868. eCollection 2025. PMID 39758967